CLINICAL TRIAL: NCT04922658
Title: A Phase II, Single-arm, Two-cohorts, Open-label, Single Center Study of Surufatinib or Surufatinib Combined With Vinorelbine as Third-line and Posterior Line Treatment in Patients With Non-Small Cell Lung Cancer
Brief Title: Surufatinib or Surufatinib Combined With Vinorelbine for Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-L106
Record Dates: First submitted 2021-06-06; First posted 2021-06-10 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — surufatinib; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surufatinib (Experimental)
  Interventions: Drug: Surufatinib
- Surufatinib plus Vinorelbine (Experimental)
  Interventions: Drug: Surufatinib Plus Vinorelbine

INTERVENTIONS:
Drug: Surufatinib — Surufatinib,300mg, qd, po, 21 days for a cycle; continuous administration until PD, death or intolerable toxicity.
  Arms: Surufatinib
Drug: Surufatinib Plus Vinorelbine — Surufatinib, 250mg, qd, po; Plus Vinorelbine, 20 mg, every 2 days; 21days for a cycle; continuous administration until PD, death or intolerable toxicity.
  Arms: Surufatinib plus Vinorelbine

SUMMARY:
A phase II study to assess the efficacy and safety of Surufatinib or Surufatinib combined with Vinorelbine as third-line and posterior line treatment in patients with NSCLC

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written Informed Consent Form (ICF) prior to any study specific procedures
2. Age ≥ 18 years, ≤80 years
3. Histologically or cytologically confirmed advanced NSCLC
4. At least two or more systemic therapies prior treatment of cytotoxic chemotherapy, treatment failure or intolerable toxicities
5. ECOG 0-2
6. Patients must have measurable lesions
7. Expected overall survival ≥6 months
8. AST, ALT and alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN)，Serum bilirubin ≤ 1.5 x ULN，creatinine<ULN
9. Prothrombin time (PT), international standard ratio (INR) ≤1.5 × ULN
10. Women of childbearing age must be willing to use adequate contraceptives during the study period of drug treatment

Exclusion Criteria:

1. Patients have received Surufatinib treatment
2. Patients with small cell lung cancer (including mixed small cell lung cancer and non-small cell lung cancer)
3. EGFR mutation /ALK rearrangement positive but not using relevant targeted drugs
4. Central squamous cell carcinoma with cavity or non-small cell lung cancer with hemoptysis (> 50 ml / D)
5. Have received other systemic anti-tumor therapies within 2 weeks before recruited(eg.chemotherapy or radiotherapy, immunotherapy, biological or hormonal therapy, or any VEGFR inhibitor treatment)
6. Participated in the clinical trials of other drugs that have not been approved or marketed in China and received the corresponding experimental drug treatment within 2 weeks before enrollment
7. systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg regardless of any antihypertensive drugs; Or patients need more than two antihypertensive drugs
8. Clinically significant electrolyte abnormality
9. Proteinuria ≥ 2+ (1.0g/24hr)
10. Patients have untreated central nervous system metastasis
11. Received any operation or invasive treatment or operation (except venous catheterization, puncture and drainage, etc.) within 4 weeks before enrollment
12. Patients have not recovered from all toxicities associated with prior anti-tumor therapy ,to acceptable baseline status, or a National Cancer Institute Common Terminology Criteria for Adverse Events(NCI CTCAE v5.0) Grade of 0 or 1, except for alopecia and oxaliplatin induced neurotoxicity ≤ 2 , and the previous surgery did not recover completely
13. Dysphagia or known malabsorption of drugs
14. Active gastric and duodenal ulcer, ulcerative colitis or uncontrolled hemorrhage in GI
15. Have evidence or history of bleeding tendency within 2 months after enrollment, the researcher assessed that moderate or severe bleeding tendency was not suitable for enrollment
16. Patients had other malignant tumors in the past 5 years or at the same time (except for the cured skin basal cell carcinoma and cervical carcinoma in situ);
17. Pregnant or lactating women
18. Allergic to Surufatinib/Vinorelbine
19. History of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation
20. Patients with acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before admission; Or a history of arterial thrombosis or deep venous thrombosis
21. There are concomitant diseases (such as severe hypertension, diabetes, thyroid disease, active infection, etc.) that seriously endanger the safety of patients or affect the completion of the study, or any laboratory abnormalities that are not suitable for participating in the clinical trial according to the judgment of the researcher
22. Serious psychological or mental disorders that may affect the compliance study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months
  To assess the efficacy of Surufatinib or Surufatinib Combined With Vinorelbine for NSCLC , patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.
Disease control rate (DCR) | up to 12 months
  CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Overall survival (OS) | up to 36 months
  The time interval between the start date of study drug and the date of death (any cause)

CONTACTS AND LOCATIONS:
Overall Officials: Yanfang Zheng, M.D., Ph.D., Principal Investigator — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No